CLINICAL TRIAL: NCT06612476
Title: Interleukin 6-guided Antibiotic Prescriptions in AECOPD Inpatients: a Multicenter Randomized Controlled Trial
Brief Title: Interleukin 6-guided Antibiotic Prescriptions in AECOPD Inpatients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-R046-02
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Chronic Obstructive Pulmonary Disease, COPD
Keywords: Aecopd; Interleukin 6; antibiotic therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interleukin 6-guided antibiotic therapy (Interleukin-6 group) (Experimental): After randomization, baseline blood samples will be drawn within 2 hours. Prescribing clinician are able to access the results of the IL-6 through the internal network of the hospital. Participants' antibiotic prescription decisions will made according to the results. The detailed recommendations are as follows: if Interleukin-6<10 pg/ml，strongly discouraged；if Interleukin-6 (10-30 pg/ml) and no sputum purulence, discouraged; if Interleukin-6 (10-30 pg/ml) and sputum purulence, Recommended; Interleukin-6>30 pg /ml, Strongly recommended.
  Interventions: Drug: Interleukin 6-guided antibiotic therapy
- GOLD-guided antibiotic therapy (GOLD group) (Active Comparator): After randomization, baseline blood samples will also need to be drawn within 2 hours. Prescribing clinician are able to access all results through the internal network of the hospital. Participants' antibiotic prescription decisions will made according to the recommendations of GOLD guideline. The guideline recommends antibiotic therapy for the following patients: those with COPD exacerbations presenting with all three cardinal symptoms (increased dyspnea, sputum volume, and sputum purulence); those with two of the cardinal symptoms, provided that increased purulence of sputum is one of them; or those who need mechanical ventilation (either invasive or noninvasive).
  Interventions: Drug: GOLD-guided antibiotic therapy

INTERVENTIONS:
Drug: Interleukin 6-guided antibiotic therapy — In Interleukin-6 group, antibiotic prescription decisions will made according to the results of IL-6.
  Arms: Interleukin 6-guided antibiotic therapy (Interleukin-6 group)
Drug: GOLD-guided antibiotic therapy — In guideline group, antibiotic prescription decisions will made according to the recommendations of GOLD guideline.
  Arms: GOLD-guided antibiotic therapy (GOLD group)

SUMMARY:
In this multicenter, prospective, randomized controlled study, we aimed to figure out, compared with the global chronic obstructive pulmonary disease initiative (GOLD) guideline -guided antibiotic therapy, whether Interleukin 6 (IL6)-guided antibiotic therapy for acute exacerbation of chronic obstructive pulmonary disease (AECOPD) can lead to a reduction in the use of antibiotics without increasing the rate of treatment failure.

DETAILED DESCRIPTION:
Acute exacerbation is the first leading cause of hospitalization and mortality among patients with COPD. Infection of bacteria has been detected in 49.59% of patients with AECOPD. Antibiotic prescriptions for AECOPD patients are usually based on GOLD guideline. However, the newest study reported that more than 85% of AECOPD inpatients received antibiotic prescription in the United States, Europe and China. Not all patients will equally experience benefit from antibiotics. Interleukin 6 (IL6) was determined as a reliable clinical biomarker in guiding antimicrobial use. It remains unclear whether IL6-guided antibiotic therapy is safe and effective for hospitalized patients with AECOPD.

The study will recruit 440 AECOPD inpatients from at least six hospitals based in China. Eligible participants will be assigned to receive either IL6-guided antibiotic therapy or GOLD-guided antibiotic therapy in 1:1 ratio randomly. The hypothesis for this study is that IL-6 guided antibiotic therapy will reduce the rate of antibiotic prescriptions for AECOPD without increasing the rate of treatment failure, compared with the group treated with GOLD-guided antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. AECOPD patients admitted to hospitals
2. The exacerbation has lasted for at least 24 hours but equal to or less than 21 days
3. ≥40 years of age but no more than 80 years old
4. With at least 10 pack-year history of smoking
5. Able to provide written informed consent and ensure the completion of the trial

Exclusion Criteria:

1. Axillary temperature≥38°C
2. Acute pneumonia identified by X-Ray or CT of the chest
3. Severe respiratory failure requiring admittance to ICU
4. Comorbidities require antibiotic therapy (i.e. infection at another site, systematic infection, active chronic inflammatory condition, specific viral infection)
5. Immunosuppression status (i.e., patients with HIV infection, with malignant tumor of blood system, receiving chemotherapy)
6. Concurrent diseases requiring corticosteroids (equivalent to 60mg prednisone/day or more than 30 days)
7. Antibiotic use in the previous four weeks
8. Current tracheotomy status
9. Bronchiectasis of origin other than COPD
10. Invasive mechanical ventilation
11. Patients diagnosed malignant tumors
12. Pregnant or lactating women, or women of childbearing age not using an acceptable method of contraception.
13. Newly diagnosed pulmonary embolism
14. Participation in another clinical trial

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of antibiotic use | During the 30-day period after randomization
  Ratio of AECOPD patients given antibiotics
Proportion of successful treatments | During the 30-day period after randomization
  Treatment success is achieved when there is a cure (full resolution of all symptoms and signs of the exacerbation) or improvement (diminishment or resolution of symptoms and signs from the exacerbation, with no additional symptoms or signs).

SECONDARY OUTCOMES:
Incidence of antibiotic use | During the first day period after randomization
  Ratio of AECOPD patients given antibiotics
Antibiotic utilization in the hospital | Between randomization and discharge, limited to 30 days
  Duration of antibiotic consumption for AECOPD and the percentage of patients treated with antibiotics for AECOPD from randomization to hospital discharge
Duration of hospitalization | Between randomization and discharge, limited to 30 days
  Total days of hospitalization until study completion, averaging 30 days
Frequency of subsequent exacerbations | During the 30-day period after randomization
  Ratio of patients who develop a subsequent acute exacerbation following recovery
Incidence of hospital readmission | Between the discharge date and 30 days post-randomization
  Ratio of patients rehospitalized for AECOPD following discharge
All-cause mortality | During the 30-day period after randomization
  Death due to any cause
Frequency of ICU admissions | During the 30-day period after randomization
  Ratio of patients admitted to the intensive care unit
noninvasive mechanical ventilation | During the 30-day period after randomization
  Ratio of patients provided with non-invasive mechanical ventilation
Change in COPD assessment test | From the initial hospital admission baseline to 30 days after randomization
  The variation from the baseline at hospital admission to 30 days after randomization
Change in St. George's Respiratory Questionnaire | From the initial hospital admission baseline to 30 days after randomization
  The variation from the baseline at hospital admission to 30 days after randomization
Change in modified Medical Research Council (mMRC) score | From the initial hospital admission baseline to 30 days after randomization
  The variation from the baseline at hospital admission to 30 days after randomization
Change in Hospital Anxiety and Depression Scale | From the initial hospital admission baseline to 30 days after randomization
  The variation from the baseline at hospital admission to 30 days after randomization

IPD SHARING:
Plan to Share IPD: No